CLINICAL TRIAL: NCT00776282
Title: An Open Label, Balanced, Randomized, Two-Treatment, Two-Sequence, Two-Period, Single-Dose, Crossover, Bioavailability Study on Loratadine Formulations Comparing Loratadine 10 mg Orally Disintegrating Tablets of Ohm Laboratories, Inc. (A Subsidiary of Ranbaxy Pharmaceuticals Inc) With Claritin® Reditabs® 10 mg Tablet (Containing Loratadine 10 mg) of Schering- Plough Healthcare Product Inc, in Healthy, Adult, Male, Human Subjects Under Fed Condition
Brief Title: Bioequivalence Study of Loratadine Orally Disintegrating Tablets 10 mg Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. tausif monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 118_LORAT_06
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: bioequivalence loratadine 10 mg orally disintegrating; tablets fed conditions
MeSH Terms: interventions — Loratadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): loratadine 10 mg orally disintegrating tablets
  Interventions: Drug: loratadine 10 mg orally disintegrating
- 2 (Active Comparator): loratadine 10 mg orally disintegrating tablets
  Interventions: Drug: loratadine 10 mg orally disintegrating

INTERVENTIONS:
Drug: loratadine 10 mg orally disintegrating

SUMMARY:
To compare the single-dose oral bioavailability of loratadine 10 mg orally disintegrating tablets of Ohm Laboratories Inc (A subsidiary of Ranbaxy Pharmaceuticals, Inc. USA) with Claritin® Reditabs® (containing loratadine 10 mg) of Schering-Plough Healthcare Product Inc., USA in healthy, adult, human male subjects under fed condition.

DETAILED DESCRIPTION:
The study was conducted as an open label, balanced, randomized, two-treatment, two-sequence,two-period, single-dose, crossover, bioavailability study on loratadine formulation comparing loratadine 10 mg orally disintegrating tablets of Ohm Laboratories, Inc. (A subsidiary of Ranbaxy pharmaceuticals Inc. USA) with Claritin® Reditabs® 10 mg Tablet (containing loratadine 10 mg) of Schering- Plough Healthcare Product Inc, USA. in healthy, adult, male, human subjects under fed condition.

A single oral dose of loratadine 10 mg orally disintegrating tablets was administered under low light condition during each period of the study under supervision of a trained medical officer.

Subjects were instructed to completely dissolve the tablet on the tongue before swallowing the saliva and then, 240 mL of water was administered 30 seconds after drug administration.

During the course of the study safety parameters assessed were vital signs, clinical examination, medical history and clinical laboratory safety tests (hematology, biochemical, serology parameters and urine analysis) at base line. Laboratory parameters of hematology and biochemistry were repeated at the end of the study.

A total of 80 subjects were randomized to receive single oral dose of Loratadine 10mg and Subjects were admitted in two groups of equal size. Group I: 1-40 Group II: 41-80 70 subjects completed both the periods of the study.

ELIGIBILITY:
Inclusion Criteria:

* Were in the age range of 18-45 years.
* Were neither overweight nor underweight for his height as per the Life Insurance Corporation of India height/weight chart for non-medical cases.
* Had voluntarily given written informed consent to participate in this study.
* Were of normal health as determined by medical history and physical examination of the subjects performed within 21 days prior to the commencement of the study.
* Had non-vegetarian dietary habit

Exclusion Criteria:

* Had history of allergy to loratadine.
* Had history of hypertension
* Had Concurrently used enzyme modifying drugs especially erythromycin, MAO inhibitors, ketoconazole, and cimetidine
* Had recent history of abdominal pain, epistaxis or sleep disturbances
* Had any evidence of organ dysfunction or any clinically significant deviation from the normal, in physical or clinical determinations.
* Had presence of disease markers of HIV 1 and 2, Hepatitis B and C viruses or syphilis infection.
* Had presence of values which were significantly different from normal reference ranges and/or judged clinically significant for haemoglobin, total white blood cells count, differential WBC count or platelet count.
* Had been positive for urinary screen testing of drugs of abuse (opiates or cannabinoids).
* Had presence of values, which are significantly different from normal reference ranges and/or judged clinically significant for serum creatinine, blood urea nitrogen, serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase, serum bilirubin, plasma glucose or serum cholesterol.
* If there was any clinically abnormal chemical and microscopic examination of urine defined as presence of RBC, WBC (>4/HPF), epithelial cells, casts, crystals, glucose (positive) or protein (positive).
* Had clinically abnormal ECG or Chest X-ray.
* Had history of serious gastrointestinal, hepatic, renal, cardiovascular, pulmonary, neurological or haematological disease, diabetes or glaucoma.
* Had history of drug dependence or excessive alcohol intake on a habitual basis of more than 2 units of alcoholic beverages per day (1 unit equivalent to half pint of beer or 1 glass of wine or 1 measure of spirit) or have difficulty in abstaining for the duration of each study period.
* Had history of any psychiatric illness, which may impair the ability to provide, written informed consent.
* Were regular smokers who smoke more than 10 cigarettes daily or have difficulty abstaining from smoking for the duration of each study period.
* Used enzyme modifying drugs within 30 days prior to Day 1 of this study.
* Had Participated in any clinical trial within 12 weeks preceding Day 1 of this study.
* Subjects who, through completion of this study, had donated and/or lost more than 350 mL of blood in the past 3 months.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2006-07; Primary Completion 2006-08 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html